CLINICAL TRIAL: NCT01371136
Title: Developing a Curriculum to Teach Laparoscopic Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Royal College of Physicians and Surgeons of Canada (Other)
Responsible Party: Principal Investigator, Teodor Grantcharov, Staff Surgeon, Unity Health Toronto
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: SMH10-059
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Education; Simulation; Technical Skills Training; Laparoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curricular Trained (Experimental): Residents in the curricular training group will participate in the entire ex-vivo training curriculum. They will train to proficiency on a virtual reality simulator. This training program has 8 tasks at an "easy", "medium" and "hard" level. They will also participate in a cognitive training component. This consists of self-directed reading, and a video training component. In the video training component, residents will watch videos of laparoscopic right and sigmoid colectomies with a staff facilitator. Finally, all residents in the intervention group will participate in a cadaver lab where they will perform a laparoscopic right or sigmoid colectomy on a cadaver.
  Interventions: Procedure: curricular training
- conventional residency training (No Intervention): These residents proceed through surgical residency training as usual

INTERVENTIONS:
Procedure: curricular training — Residents in the curricular training group will participate in the entire ex-vivo training curriculum. They will train to proficiency on a virtual reality simulator. This training program has 8 tasks at an "easy", "medium" and "hard" level. They will also participate in a cognitive training component. This consists of self-directed reading, and a video training component. In the video training component, residents will watch videos of laparoscopic right and sigmoid colectomies with a staff facilitator. Finally, all residents in the intervention group will participate in a cadaver lab where they will perform a laparoscopic right or sigmoid colectomy on a cadaver.
  Arms: Curricular Trained

SUMMARY:
Although a significant amount of work has been done to validate simulators as viable systems to teach technical skills outside the operating room, the next necessary step is to integrate simulator training into a comprehensive curriculum. The purpose of this study is to develop and validate a comprehensive ex-vivo curriculum for laparoscopic colorectal surgery. This curriculum will include training on a virtual reality simulator, cognitive training and cadaver lab training. The investigators will assess the effectiveness of the curriculum by conducting a randomized single blinded controlled trial. The investigators will be comparing the technical performance of curricular trained and non-trained residents in the operating room, during a procedure on a patient. The investigators hypothesize that surgical residents who participate in the curriculum will have superior technical proficiency and cognitive knowledge relating to performing laparoscopic colorectal surgery compared to conventionally trained residents.

ELIGIBILITY:
Inclusion Criteria:

* resident in general surgery
* post graduate year (PGY) 2 or higher
* performed less than 10 laparoscopic colorectal procedures independently

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Difference in operating room performance between intervention and control group | 5 months from intervention
  Surgical residents participating in the study will perform a laparoscopic right colectomy in the operating room. The procedure will be video-recorded through the laparoscopic camera. The videos will be given to a blinded expert in video assessment who will assess the technical proficiency of the resident using a validated global rating scale.

SECONDARY OUTCOMES:
Difference in cognitive knowledge between intervention and control group | 5 months from the intervention
  Residents in both groups will complete a multiple choice test designed to assess the amount of cognitive knowledge they have relating to the technical steps of performing laparoscopic colorectal surgery
Difference in technical performance on the virtual reality simulator between intervention and control group residents | 5 months from intervention
  Study participants will complete the easy level of the virtual reality training portion of the curriculum

CONTACTS AND LOCATIONS:
Overall Officials: Teodor P Grantcharov, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Palter VN, Grantcharov TP. Development and validation of a comprehensive curriculum to teach an advanced minimally invasive procedure: a randomized controlled trial. Ann Surg. 2012 Jul;256(1):25-32. doi: 10.1097/SLA.0b013e318258f5aa. PMID 22664557